CLINICAL TRIAL: NCT02539563
Title: Do Peanut Shaped Birthing Balls Reduce the Length of Labor in Patients With Epidural Analgesia?
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: During interim analysis, it appeared there were no difference in groups
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: IRB00033103
Record Dates: First submitted 2015-08-25; First posted 2015-09-03 (Estimated); Results first posted 2019-04-29 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2018-07

CONDITIONS: Labor
Keywords: labor duration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- peanut ball (Active Comparator): the peanut shaped birthing ball after labor analgesia will be utilized
  Interventions: Other: peanut shaped birthing ball
- no peanut ball (No Intervention): the peanut shaped birthing ball will not be utilized during labor

INTERVENTIONS:
Other: peanut shaped birthing ball — peanut ball will be utilized
  Arms: peanut ball

SUMMARY:
Labor patients who meet inclusion and exclusion criteria will be consented to be participate in this study to determine if the use of a peanut shaped birthing ball reduces the length of labor and reduces the incidence of cesarean section. Subjects will be randomized at the time of consent to either use the birthing ball or not use the birthing ball from the time of labor analgesia until complete cervical dilation.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous
* >/= 18 years of age
* not allergic to medications used for labor analgesia
* no contraindications to labor analgesia
* ASA I-II
* EGA >/= 37 weeks

Exclusion Criteria:

* under age 18
* Spanish speaking only
* multiparous
* EGA <37 weeks

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 101 (Actual)
Dates: Start 2015-06-04 (Actual); Primary Completion 2017-12-26 (Actual); Study Completion 2017-12-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert D'Angelo, MD, Principal Investigator — WakeForest School of Medicine
Locations (1):
- Novant Health-Forsyth Medical Center, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bucklin BA, Hawkins JL, Anderson JR, Ullrich FA. Obstetric anesthesia workforce survey: twenty-year update. Anesthesiology. 2005 Sep;103(3):645-53. doi: 10.1097/00000542-200509000-00030. No abstract available. PMID 16129992
- [Background] Halpern SH, Leighton BL, Ohlsson A, Barrett JF, Rice A. Effect of epidural vs parenteral opioid analgesia on the progress of labor: a meta-analysis. JAMA. 1998 Dec 23-30;280(24):2105-10. doi: 10.1001/jama.280.24.2105. PMID 9875879
- [Background] Martin JA, Hamilton BE, Osterman MJ, Curtin SC, Matthews TJ. Births: final data for 2013. Natl Vital Stat Rep. 2015 Jan 15;64(1):1-65. PMID 25603115
- [Background] American College of Obstetricians and Gynecologists (College); Society for Maternal-Fetal Medicine; Caughey AB, Cahill AG, Guise JM, Rouse DJ. Safe prevention of the primary cesarean delivery. Am J Obstet Gynecol. 2014 Mar;210(3):179-93. doi: 10.1016/j.ajog.2014.01.026. PMID 24565430
- [Background] Tussey CM, Botsios E, Gerkin RD, Kelly LA, Gamez J, Mensik J. Reducing Length of Labor and Cesarean Surgery Rate Using a Peanut Ball for Women Laboring With an Epidural. J Perinat Educ. 2015;24(1):16-24. doi: 10.1891/1058-1243.24.1.16. PMID 26937158
- [Background] Tsen LC, Thue B, Datta S, Segal S. Is combined spinal-epidural analgesia associated with more rapid cervical dilation in nulliparous patients when compared with conventional epidural analgesia? Anesthesiology. 1999 Oct;91(4):920-5. doi: 10.1097/00000542-199910000-00010. PMID 10519493
- [Background] BISHOP EH. PELVIC SCORING FOR ELECTIVE INDUCTION. Obstet Gynecol. 1964 Aug;24:266-8. No abstract available. PMID 14199536

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Peanut Ball | no Peanut Ball
Started | 45 | 56
Completed | 39 | 42
Not Completed | 6 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Peanut Ball | no Peanut Ball | Total
Number analyzed (Participants) | 39 | 42 | 81
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 39 | 42 | 81
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 39 | 42 | 81
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 7 | 11 | 18
  White | 32 | 30 | 62
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 39 | 42 | 81
Height [Mean (Standard Deviation); unit: centimeters] — Population: analysis performed on those completing study only
  centimeters | 165.1 (5.1) | 161.3 (7.6) | 163.2 (6.4)
Weight [Mean (Standard Deviation); unit: kilograms] — Population: analysis performed on those completing study only
  kilograms | 91.4 (21.4) | 90.5 (22.7) | 90.9 (21.9)
Gestational Age [Mean (Standard Deviation); unit: weeks] | 39.5 (1.23) | 39.6 (1.31) | 39.55 (1.27)
Oxytocin Augmentation [Count of Participants; unit: Participants] — those receiving oxytocin in order for labor to be augmented
  Participants | 24 | 28 | 52

OUTCOME MEASURES:

1. Primary Outcome: Length of Labor
Description: time in minutes will be calculated from epidural catheter insertion until delivery
Time Frame: up to 24 hours
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Peanut Ball | no Peanut Ball
Number analyzed (Participants) | 39 | 42
minutes | 387 (256) | 441 (269)

2. Secondary Outcome: Maternal Satisfaction
Description: 11-point scale of 0=not satisfied up to 10=most satisfied of all
Time Frame: length of labor, up to 24 hours
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Peanut Ball | no Peanut Ball
Number analyzed (Participants) | 39 | 42
units on a scale | 8.86 (2.01) | 7.88 (2.68)

3. Secondary Outcome: Participant Cesarean Delivery Incidence-Mode of Deliveries
Description: the number of subjects who had to had a cesarean delivery
Time Frame: up to 24 hours
Measure: Number; unit: number of cesarean deliveries
Arm/Group | Peanut Ball | no Peanut Ball
Number analyzed (Participants) | 39 | 42
number of cesarean deliveries | 15 | 15

4. Secondary Outcome: Number of Participants With Post-delivery Complications
Description: Number of participants that had post-delivery complications was reported
Time Frame: up to 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Peanut Ball | no Peanut Ball
Number analyzed (Participants) | 39 | 42
Participants | 0 | 0

5. Post Hoc Outcome: Cervical Dilation
Description: rate in centimeters per hour of dilation
Time Frame: length of labor, up to 24 hours
Population: rate of cervical dilation in centimeters per hour that subjects dilated in each group
Measure: Mean (Standard Deviation); unit: centimeters per hour
Arm/Group | Peanut Ball | no Peanut Ball
Number analyzed (Participants) | 39 | 42
centimeters per hour | 1.49 (0.95) | 1.74 (2.37)

ADVERSE EVENTS:
Time Frame: thoughout the length of labor
Arm/Group | Peanut Ball | no Peanut Ball
All-Cause Mortality (participants affected / at risk) | 0/39 | 0/42
Serious Adverse Events (participants affected / at risk) | 0/39 | 0/42
Other Adverse Events (participants affected / at risk) | 0/39 | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-01): https://cdn.clinicaltrials.gov/large-docs/63/NCT02539563/Prot_SAP_000.pdf